CLINICAL TRIAL: NCT04192695
Title: Surveillance and Early Detection of Esophageal Squamous Cell Carcinoma With Minimally-invasive Cytosponge™ Cell Collection Device Coupled With Molecular Biomarkers
Brief Title: Esophageal Squamous Cell Cancer Surveillance With Cytosponge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Wladyslaw Januszewicz, Principal Investigator, Centre of Postgraduate Medical Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 109/PB/2019
Record Dates: First submitted 2019-11-12; First posted 2019-12-10 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Gastroscopy; Biopsy

STUDY DESIGN:
Intervention Model Description: A prospective cohort study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cytosponge (Experimental): This part of the study will have an active prospective recruitment of patients. Recruitment will involve two patient populations:
  1. Patients with ESCC
  2. Patients at high risk for ESCC
  Following inclusion in the study, subjects will be asked to complete a behavior questionnaire, have blood collected, and undergo a Cytosponge™ procedure followed by diagnostic gastroscopy using advanced imaging with biopsies. During gastroscopy, additional tissue samples will be collected for research purposes. These samples, along with cytological specimens from the Cytosponge™, will be analyzed to assess the diagnostic accuracy of biomarkers in the diagnosis of LG-IEN, HG-IEN, and ESCC.
  Interventions: Device: Cytosponge cell collection device

INTERVENTIONS:
Device: Cytosponge cell collection device — The Cytosponge™ is a minimally-invasive sampling device consisting of a polyurethane sponge compressed in a cellophane capsule attached to a string. When swallowed, the capsule dissolves in the stomach, releasing the cell collection sponge that expands to 3 cm in diameter. Next, a nurse or qualified medical technician retrieves the sponge by pulling back on the string and retracting it through the mouth. During extraction, the rough texture on the surface of the sponge collects epithelial cells in the cardia and along the entire length of the esophagus. Cytosponge™ has excellent safety profile and is approved by the Food and Drug Administration (FDA) and the Healthcare Products Regulatory Agency (HPRA) in the UK.
  Other Names: Gastroscopy with biopsies

SUMMARY:
Surveillance and early detection of esophageal squamous cell carcinoma with minimally-invasive Cytosponge™ cell collection device coupled with molecular biomarkers.

DETAILED DESCRIPTION:
The goal of the study is to identify molecular abnormalities at each developmental stage of esophageal squamous cell carcinoma (low-grade intraepithelial neoplasia, high-grade intraepithelial neoplasia, and early squamous cell carcinoma) in order to establish new molecular biomarkers with potential for early detection and surveillance of the disease using the minimally-invasive Cytosponge™ cell collection device. Firstly, tissue samples after endoscopic treatment (endoscopic mucosal resection and endoscopic submucosal dissection) for squamous intraepithelial neoplasia and early squamous cell carcinoma will be analyzed with the use of the next-generation sequencing to identify potential diagnostic biomarkers. Afterward, patients with- and at risk- of esophageal squamous cell carcinoma will be recruited to undergo a diagnostic endoscopy with biopsies (the gold standard) and Cytosponge procedure. The diagnostic accuracy of Cytosponge coupled with molecular biomarkers will be evaluated to compare with the gold standard.

ELIGIBILITY:
Inclusion Criteria:

Patients with esophageal squamous cell cancer (ESCC):

* Patients ≥18 years of with adequate performance status for endoscopy
* Newly diagnosed ESCC suitable for endoscopic or oncological treatment (Rth/Chth)
* Patients currently undergoing oncological treatment (Rth/Chth)
* Consent to provide tissue samples for the study
* Dysphagia grade ≤2 (able to swallow mixed foods and tablets)

Patients at high risk for ESCC:

* Patients ≥18 years of age with adequate performance status for endoscopy
* Prior definitive treatment for head and neck cancer (cancer of the oral cavity, hypopharyngeal cancer, laryngeal carcinoma) and at least 12 months post-therapy (both Rth, Chth, and combination treatment)
* Prior definitive endoscopic treatment for early ESCC in the past (at least 6 months since completion)
* Consent to provide tissue samples for the study
* Dysphagia grade ≤2

Exclusion Criteria (for both groups of patients):

* Patients currently on anticoagulant treatment (warfarin, acenocoumarol) with no possibility of stopping / modification
* Dysphagia grade ≥3 (able to swallow only liquid foods)
* History of myocardial infarction or other cardiovascular event within 6 months of enrolment
* Neurological diseases associated with impaired swallowing
* Patients in long-term care or institutional care (physical, psycho-social disorders, intellectual disability).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Discovery of suitable biomarkers for squamous intraepithelial neoplasia to inform future trials. | 4 years
  RNA-seq expression analysis will be used to measure the abundance of the previously identified biomarkers of squamous intraepithelial neoplasia, including genes TP53, NFE2L2, MLL2, ZNF750, NOTCH1, TFNAIP3, and CHN1. The study will include these biomarkers, but will not be limited to them.

SECONDARY OUTCOMES:
Acceptability of the Cytosponge™ cell collection device in patients with ESCC and high-risk for ESCC | 4 years
  % of Participants that have scored the Cytosponge experience of at least 6 points on a 0 to 10 Visual Analogue Scale (VAS) acceptability scale whereby 0 denotes "worst experience in life" and 10 denotes "best experience in life".
Safety of the Cytosponge™ cell collection device in patients with ESCC and high-risk for ESCC: rate of Participants with adverse events within 30 days after application | 4 years
  The rate of Participants with adverse events within 30 days after application of the Cytosponge cell collection device, which is defined as any event that require admission to the hospital. E.g. retention of the device in the GI tract, chest pain or gastrointestinal bleeding requiring admission to the Ward

CONTACTS AND LOCATIONS:
Overall Officials: Wladyslaw Januszewicz, M.D., Principal Investigator — Centre of Postgraduate Medical Education, Warsaw, Poland
Locations (1):
- Medical Centre for Postgraduate Education, Warsaw, Poland

REFERENCES:
- [Derived] Turkot MH, Yusuf A, Nowicki-Osuch K, Pilonis ND, Malhotra S, O'Donovan M, Mroz A, Lenarcik M, Wronska E, Mikula M, Zwolinski J, Wojtowicz-Popiel M, di Pietro M, Regula J, Kaminski MF, Fitzgerald RC, Januszewicz W. Feasibility and diagnostic accuracy of a capsule-sponge device for esophageal squamous neoplasia (EDEN trial). Clin Gastroenterol Hepatol. 2026 Jan 31:S1542-3565(26)00053-4. doi: 10.1016/j.cgh.2026.01.025. Online ahead of print. PMID 41628756